CLINICAL TRIAL: NCT04566757
Title: Safety and Efficacy of Human Umbilical Cord Blood Plasma Infusion for Age-Related Cognitive Decline
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: American Academy of Regenerative Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AARM2020
Record Dates: First submitted 2020-09-04; First posted 2020-09-28 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Age-related Cognitive Decline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Umbilical Cord Plasma Infusion (Experimental): Infusion of 50cc of Umbilical Cord Blood Plasma bi-monthly for 6 months
  Interventions: Biological: Umbilical Cord Blood Plasma

INTERVENTIONS:
Biological: Umbilical Cord Blood Plasma — Intravenous Infusion of Umbilical Cord Blood Plasma

SUMMARY:
This study is designed to investigate the safety of Umbilical Cord Blood Plasma infusions in elderly adults regardless of gender, with age-related cognitive decline. Human clinical data of the use of young plasma appear to show beneficial cognitive effects.

ELIGIBILITY:
Inclusion Criteria:

1. Age 65-85 years old
2. Evidence of cognitive decline on neuro-cognitive testing
3. Able to participate in research trial for 12 months
4. Women must have documented menopause or infertility determination
5. Ability to receive intravenous infusions
6. Patient or legally authorized representative able to sign informed consent

Exclusion Criteria:

1. Patients receiving any other investigational biologics or drugs
2. History of transfusion reaction
3. Dementia related to specific pathology (Alzheimer's Disease, Alcohol-related, etc.)
4. Inability to participate in cognitive or performance testing
5. History of cancer in the last 5 years
6. History of infectious disease within the previous 12 months
7. Severe kidney (eGFR< 30) and heart failure (Class III/IV)
8. History of Human Immunodeficiency Virus Infection
9. History of Hepatitis B, or C
10. History of immunosuppressive therapy
11. History of organ transplantation
12. Difficulty of obtaining peripheral venous access
13. Allergy to histamine blockers
14. Inability to participate in the clinical trial at any data collection and end points

    -

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-06-14 (Estimated)

PRIMARY OUTCOMES:
Safety of Umbilical Cord Blood Plasma Infusion | 6 months
  Assessment of Human Leukocyte Antigen (HLA) in recipient following Umbilical Cord Blood Plasma infusion

SECONDARY OUTCOMES:
Assessment of Executive Function | 12 months
  Assessment of executive function by Wisconsin Card Sorting Test (WCST)
Assessment of Working Memory | 12 months
  Assessment of working memory by Wechsler Memory Scale

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Horowitz AM, Villeda SA. Therapeutic potential of systemic brain rejuvenation strategies for neurodegenerative disease. F1000Res. 2017 Aug 1;6:1291. doi: 10.12688/f1000research.11437.1. eCollection 2017. PMID 28815019
- [Background] Villeda SA, Luo J, Mosher KI, Zou B, Britschgi M, Bieri G, Stan TM, Fainberg N, Ding Z, Eggel A, Lucin KM, Czirr E, Park JS, Couillard-Despres S, Aigner L, Li G, Peskind ER, Kaye JA, Quinn JF, Galasko DR, Xie XS, Rando TA, Wyss-Coray T. The ageing systemic milieu negatively regulates neurogenesis and cognitive function. Nature. 2011 Aug 31;477(7362):90-4. doi: 10.1038/nature10357. PMID 21886162
- [Background] Kang S, Moser VA, Svendsen CN, Goodridge HS. Rejuvenating the blood and bone marrow to slow aging-associated cognitive decline and Alzheimer's disease. Commun Biol. 2020 Feb 13;3(1):69. doi: 10.1038/s42003-020-0797-4. PMID 32054965
- [Background] Villeda SA, Plambeck KE, Middeldorp J, Castellano JM, Mosher KI, Luo J, Smith LK, Bieri G, Lin K, Berdnik D, Wabl R, Udeochu J, Wheatley EG, Zou B, Simmons DA, Xie XS, Longo FM, Wyss-Coray T. Young blood reverses age-related impairments in cognitive function and synaptic plasticity in mice. Nat Med. 2014 Jun;20(6):659-63. doi: 10.1038/nm.3569. Epub 2014 May 4. PMID 24793238